CLINICAL TRIAL: NCT05805033
Title: Peri-Implant Soft Tissue Integration in Humans: Influence of Material
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Clémentine CANUEL, 2nd year resident in periodontology, oral and implant surgery, Centre Hospitalier Universitaire de Liege
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022/189; B7072022000023 (Other: Comité de étique Hospitalo-Facultaire Universitaire de Liege)
Record Dates: First submitted 2023-03-28; First posted 2023-04-07 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ultra-polished zirconia abutment (Experimental)
  Interventions: Other: Mucointegration
- Machined zirconia abutment (Experimental)
  Interventions: Other: Mucointegration
- Titanium abutment (Active Comparator)
  Interventions: Other: Mucointegration

INTERVENTIONS:
Other: Mucointegration — Placement of abutment on a dental implant to study mucointegration

SUMMARY:
The purpose of this study is to compare the mucointegration of 2 types of surface roughness of zirconia abutments with titanium. The surface roughness will be machined and ultra-polished.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants give written informed consent and eligibility for study entry.

The day of the surgery, patients will be randomized in machined zirconia or ultra-polished zirconia.

After 8 weeks of healing, biopsy are separated in two groups according to the removal:

* if the abutment come together with the surrounding soft tissues, it goes for a non decalcified histology for histometric measurements to determine the dimensions of biological width (sulcus depth, epithelial and connective adhesion)
* if the abutment come separate of the surrounding tissue, the soft tissue goes for immunohistochemistry to analyse pro-inflammatory cells and vascularisation and the abutment for SEM analysis to calculate the percentage of adhesion of the cells on the abutment

ELIGIBILITY:
Inclusion Criteria:

* Participants have to voluntarily sign the informed consent form before any study related action
* Patients aged 18 or over
* Patients with one or more missing teeth in the maxillary or mandible area, seeking implant therapy
* Men/women
* Patients in good systemic health (ASA I/ II) and no contraindication for oral surgical interventions
* Patients requiring a replacement of missing teeth; the tooth at the implant site(s) must have been extracted or lost at least 12 weeks before the date of implantation
* At least 3 mm of fibrous mucosa in the bucco-lingual dimension
* Full mouth plaque score (FMPI) lower than or equal to 25%
* At least a diameter of 4 mm for the implant (regular diameter)

Exclusion Criteria:

* Autoimmune disease requiring medical treatment
* Medical conditions requiring prolonged use of steroids
* Use of Bisphosphonates intravenously or more than 3 years of oral use
* Infection (local or systemic) - patients with gingivitis or active local infection will undergo a medical treatment prior to the entrance to the study, and each individual will be evaluated for suitability; in case of a systemic infection, the evaluation will be based on medical anamneses, and if necessary, a patient will be referred to relevant medical tests
* Current pregnancy or breastfeeding women
* Alcoholism or chronical drug abuse
* Immunocompromised patients
* Uncontrolled diabetes
* Smokers
* Prisoners
* Implant's diameter under 4 mm (narrow implant)
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of the study or interference with analysis of study results, such as history of non-compliance, or unreliability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Histomorphometry | 8 weeks of healing
  Height measure of biological width (sulcus depth, epithelial and connective adhesion)
Immunohistology | 8 weeks of healing
  Analysis of the pro-inflammatory cells and vascularisation of the soft tissue + analysis of the percentage of cells adhesion on the abutment

CONTACTS AND LOCATIONS:
Locations (1):
- Clémentine Canuel, Liège, Belgium